CLINICAL TRIAL: NCT04436276
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2a Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Ad26COVS1 in Adults Aged 18 to 55 Years Inclusive and Adults Aged 65 Years and Older
Brief Title: A Study of Ad26.COV2.S in Adults (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR108828; 2020-001483-28 (EudraCT Number); VAC31518COV1001 (Other: Janssen Vaccines & Prevention B.V.)
Expanded Access: NCT04817657 (No longer available)
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Covid-19 Prevention
Keywords: COVID-19; Ad26COVS1; Ad26.COV2.S; SARS CoV 2; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1a (Experimental): Participants (healthy adults aged greater than or equal to (>=)18 to less than or equal to (<=) 55 years) will receive Ad26.COV2.S at 2 dose levels, as a single dose or 2 dose schedule with an 8-week interval or matching Placebo on Day 1 and Day 57. At unblinding visit, post Emergency Use Authorization (EUA), conditional licensure, or approval for the single dose regimen of Ad26.COV2.S vaccine, participants initially receiving placebo will be offered to receive a single dose of Ad26.COV2.S. If they choose not to receive Ad26.COV2.S they will be asked to continue to be followed in this study. All eligible participants who have previously received coronavirus disease-2019 (COVID-19) vaccination (as primary regimen or additional dose) if the last vaccination was >=6 months ago, will be offered to receive a single ad hoc booster dose of Ad26.COV2.S. If they choose not to receive ad-hoc booster dose they will be asked to continue to be followed in this study.
  Interventions: Biological: Ad26.COV2.S; Biological: Placebo
- Cohort 1b (Experimental): Participants (healthy adults aged >=18 to <= 55 years) will receive Ad26.COV2.S as a single vaccination in the primary regimen or matching Placebo on Day 1 and Day 57. At unblinding visit, post EUA, conditional licensure, or approval for the single dose regimen of Ad26.COV2.S vaccine, participants initially receiving placebo will be offered to receive a single dose of Ad26.COV2.S. If they choose not to receive Ad26.COV2.S they will be asked to continue to be followed in this study. All eligible participants who have previously received any COVID-19 vaccination (as primary regimen or additional dose) if the last vaccination was >=6 months ago will be offered to receive a single ad hoc booster dose of Ad26.COV2.S. If they choose not to receive ad-hoc booster dose they will be asked to continue to be followed in this study.
  Interventions: Biological: Ad26.COV2.S; Biological: Placebo
- Cohort 2a (Experimental): Participants (healthy adults aged >=18 to <=55 years) will receive Ad26.COV2.S as single vaccination in the primary regimen or matching Placebo on Day 1, followed by booster vaccination at 6 or 12 months with same dose or matching Placebo. At unblinding visit, post EUA, conditional licensure, or approval for the single dose regimen of Ad26.COV2.S vaccine, participants initially receiving placebo will be offered to receive a single dose of Ad26.COV2.S vaccine and who are not willing to receive single dose of Ad26.COV2.S vaccine will continue to receive booster vaccination. All eligible participants who have previously received any COVID-19 vaccination (as primary regimen or additional dose) if the last vaccination was >= 6 months ago, will be offered to receive a single ad hoc booster dose of Ad26.COV2.S and who are not willing to receive single ad hoc booster dose of Ad26.COV2.S or are not eligible to receive the ad hoc booster dose will continue to receive booster vaccination.
  Interventions: Biological: Ad26.COV2.S; Biological: Placebo
- Cohort 2b (Experimental): Participants(healthy adults aged >=18 to <=55 years)will receive Ad26.COV2.S in primary regimen or matching Placebo on Day 1 and 57,followed by booster vaccination at 8 or 14 months (that is, 6 or 12 months after completion of primary regimen)with same dose or matching Placebo.At unblinding visit,post EUA,conditional licensure,or approval for single dose regimen of Ad26.COV2.S vaccine,participants initially receiving placebo will be offered to receive single dose of Ad26.COV2.S vaccine and who are not willing to receive single dose of Ad26.COV2.S vaccine will continue to receive booster vaccination.All eligible participants who have previously received any COVID-19 vaccination(as primary regimen or additional dose)if last vaccination was >= 6 months ago,will be offered to receive single ad hoc booster dose of Ad26.COV2.S and who are not willing to receive single ad hoc booster dose of Ad26.COV2.S or are not eligible for ad hoc booster dose will continue to receive booster vaccination.
  Interventions: Biological: Ad26.COV2.S; Biological: Placebo
- Cohort 3 (Experimental): Participants (good or stable health adults aged >=65 years) will receive Ad26.COV2.S at 2 dose levels, as a single dose or 2 dose schedule with an 8-week interval or matching Placebo on Day 1 and Day 57. At unblinding visit, post EUA, conditional licensure, or approval for the single dose regimen of Ad26.COV2.S vaccine, participants initially receiving placebo will be offered to receive a single dose of Ad26.COV2.S. If they choose not to receive Ad26.COV2.S they will be asked to continue to be followed in this study. All eligible participants who have previously received any COVID-19 vaccination (as primary regimen or additional dose) if the last vaccination was >=6 months ago will be offered to receive a single ad hoc booster dose of Ad26.COV2.S. If they choose not to receive ad-hoc booster dose or if they are not eligible for ad-hoc booster dose, then they will be asked to continue to be followed in this study.
  Interventions: Biological: Ad26.COV2.S; Biological: Placebo

INTERVENTIONS:
Biological: Ad26.COV2.S — Participants will receive intramuscular (IM) injection of Ad26.COV2.S.
  Other Names: JNJ-78436735; Ad26COVS1
Biological: Placebo — Participants will receive Placebo.

SUMMARY:
The purpose of the study is to assess the safety, reactogenicity, and immunogenicity of Ad26.COV2.S at 2 dose levels, administered intramuscularly (IM) as a single-dose or 2-dose schedule, with a single booster vaccination administered in one cohort in healthy adults aged greater than or equal to (>=) 18 to less than or equal to (<=) 55 years and in adults aged >= 65 years in good health with or without stable underlying conditions. The purpose of the study is also to assess the safety and reactogenicity of Ad26.COV2.S administered as ad hoc booster vaccination in healthy adults aged >= 18 to <= 55 years and in adults >= 65 years in good health with or without stable underlying conditions.

ELIGIBILITY:
Inclusion criteria:

* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose, procedures, and potential risks and benefits of the study, and is willing to participate in the study
* All female participants of childbearing potential must have a negative highly sensitive urine pregnancy test at screening; and have a negative highly sensitive urine pregnancy test immediately prior to each study vaccine administration
* Participant must have a body mass index (BMI) less than or equal to (<=) 30.0 kilograms per square meter (kg/m^2)
* Applicable to Cohorts 1 and 2 only: Participant must be healthy, in the investigator's clinical judgment, as confirmed by medical history, physical examination, clinical laboratory assessments, and vital signs performed at screening, and must not have comorbidities related to an increased risk of severe coronavirus disease-2019 (COVID-19). Applicable to Cohort 3 only: In the investigator's clinical judgment, participant must be either in good or stable health Participants may have underlying illnesses such as hyperlipoproteinemia or hypothyroidism, as long as their symptoms and signs are medically controlled and not considered to be comorbidities related to an increased risk of severe COVID-19 (participants may have medical conditions of mild severity (according to the Toxicity Grading Scale), as long as it is stable and medically controlled as defined by no change in medication over the past 6 months (except for issues of tolerability or use of similar drug with same mechanism of action, for example, thiazides, Beta blockers, Alpha blockers at the same effective dose).

Exclusion criteria:

* Participant has a clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature greater than or equal to (>=) 38.0 degree Celsius within 24 hours prior to the planned first dose of study vaccine; randomization at a later date is permitted at the discretion of the investigator and after consultation with the sponsor
* Participant has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has a history of any neurological disorders or seizures including Guillain-Barre syndrome, with the exception of febrile seizures during childhood
* Participant has a positive diagnostic test result for SARS-CoV-2 infection confirmed by polymerase chain reaction (PCR) at screening
* Participants with comorbidities that are or might be associated with an increased risk of progression to severe COVID-19, that is, participants with moderate-to-severe asthma; chronic lung diseases such as chronic obstructive pulmonary disease (COPD) (including emphysema and chronic bronchitis), idiopathic pulmonary fibrosis and cystic fibrosis; diabetes (including type 1 or type 2); serious heart conditions, including heart failure, coronary artery disease, congenital heart disease, cardiomyopathies, and (pulmonary) hypertension or high blood pressure; obesity (BMI >= 30 kg/m^2); chronic liver disease, including cirrhosis; sickle cell disease; thalassemia; cerebrovascular disease; neurologic conditions (dementia); smoking end stage renal disease; organ transplantation; cancer; HIV infection and other immunodeficiencies; hepatitis B infection; and sleep apnea. Applicable to Cohort 3 only: Participants may have hypertension of mild severity (according to the Toxicity Grading Scale), as long as it is stable and medically controlled as defined by no change in medication over the past 6 months (except for issues of tolerability or use of similar drug with same mechanism of action, for example, thiazides, Beta blockers, Alpha blockers at the same effective dose)
* Applicable to Cohorts 1 and 3 only: Participant currently working in an occupation with a high risk of exposure to SARS-CoV-2 (for example, health care worker or emergency response personnel) or considered at the investigator's discretion to be at increased risk to acquire COVID-19 for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (12):
- United States (7):
  - Optimal Research, San Diego, California
  - Optimal Research, Melbourne, Florida
  - Optimal Research, Peoria, Illinois
  - Optimal Research, Rockville, Maryland
  - Center for Virology and Vaccine Research, Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee
  - Optimal Research, Austin, Texas
- Belgium (5):
  - Universiteit Antwerpen - Centrum voor de Evaluatie van Vaccinaties (CEV), Edegem
  - UZA-SGS, Edegem
  - Center for Vaccinology (CEVAC), Ghent
  - UZ Leuven, Leuven
  - Clinical Pharmacology Unit, Merksem

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Sadoff J, Le Gars M, Brandenburg B, Cardenas V, Shukarev G, Vaissiere N, Heerwegh D, Truyers C, de Groot AM, Jongeneelen M, Kaszas K, Tolboom J, Scheper G, Hendriks J, Ruiz-Guinazu J, Struyf F, Van Hoof J, Douoguih M, Schuitemaker H. Durable antibody responses elicited by 1 dose of Ad26.COV2.S and substantial increase after boosting: 2 randomized clinical trials. Vaccine. 2022 Jul 30;40(32):4403-4411. doi: 10.1016/j.vaccine.2022.05.047. Epub 2022 Jun 3. PMID 35667914
- [Derived] Stephenson KE, Le Gars M, Sadoff J, de Groot AM, Heerwegh D, Truyers C, Atyeo C, Loos C, Chandrashekar A, McMahan K, Tostanoski LH, Yu J, Gebre MS, Jacob-Dolan C, Li Z, Patel S, Peter L, Liu J, Borducchi EN, Nkolola JP, Souza M, Tan CS, Zash R, Julg B, Nathavitharana RR, Shapiro RL, Azim AA, Alonso CD, Jaegle K, Ansel JL, Kanjilal DG, Guiney CJ, Bradshaw C, Tyler A, Makoni T, Yanosick KE, Seaman MS, Lauffenburger DA, Alter G, Struyf F, Douoguih M, Van Hoof J, Schuitemaker H, Barouch DH. Immunogenicity of the Ad26.COV2.S Vaccine for COVID-19. JAMA. 2021 Apr 20;325(15):1535-1544. doi: 10.1001/jama.2021.3645. PMID 33704352
- [Derived] Sadoff J, Le Gars M, Shukarev G, Heerwegh D, Truyers C, de Groot AM, Stoop J, Tete S, Van Damme W, Leroux-Roels I, Berghmans PJ, Kimmel M, Van Damme P, de Hoon J, Smith W, Stephenson KE, De Rosa SC, Cohen KW, McElrath MJ, Cormier E, Scheper G, Barouch DH, Hendriks J, Struyf F, Douoguih M, Van Hoof J, Schuitemaker H. Interim Results of a Phase 1-2a Trial of Ad26.COV2.S Covid-19 Vaccine. N Engl J Med. 2021 May 13;384(19):1824-1835. doi: 10.1056/NEJMoa2034201. Epub 2021 Jan 13. PMID 33440088
- [Derived] Bos R, Rutten L, van der Lubbe JEM, Bakkers MJG, Hardenberg G, Wegmann F, Zuijdgeest D, de Wilde AH, Koornneef A, Verwilligen A, van Manen D, Kwaks T, Vogels R, Dalebout TJ, Myeni SK, Kikkert M, Snijder EJ, Li Z, Barouch DH, Vellinga J, Langedijk JPM, Zahn RC, Custers J, Schuitemaker H. Ad26 vector-based COVID-19 vaccine encoding a prefusion-stabilized SARS-CoV-2 Spike immunogen induces potent humoral and cellular immune responses. NPJ Vaccines. 2020 Sep 28;5:91. doi: 10.1038/s41541-020-00243-x. eCollection 2020. PMID 33083026

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1085 participants were enrolled in the study, out of which 1076 participants received treatment. Remaining 9 participants did not receive any treatment and are excluded from the analyses.
Groups:
- COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10): Healthy adult participants aged greater than or equal to (>=) 18 to less than or equal to (<=) 55 received a single intramuscular (IM) injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad hoc booster vaccination (AHBV) of Ad26.COV2.S at the dose of 5*10^10 >=6 months after Vaccination 2.
- COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and matching placebo (PL) on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10); COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10); COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and matching placebo on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 1A: Placebo, Placebo; COHORT 1B: Placebo, Placebo: Healthy adult participants aged >=18 to <=55 received a single IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1 (vaccination1) and 57 (Vaccination2). As per protocol amendment 10, after unblinding, enrolled participants who had initially received placebo were offered a single dose of 5*10^10 vp Ad26.COV2.S.
- COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and a matching placebo on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10): Group 1 and Group 4 healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) followed by matching placebo at 6 and 12 months as matching Booster (B) 1 and Booster 2 vaccination. As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S. 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL: Group 2 healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) followed by first booster vaccination with single IM injection of Ad26.COV2.S 5*10^10 vp booster 1 at 6 months and a matching placebo at 12 months to match second Booster vaccination.
- COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10: Group 3 healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) followed by a matching placebo booster 1 injection after 6 months and Ad26.COV2.S 5*10^10 vp after 12 months as Booster 2.
- COHORT 2A: Placebo, B: PL: Group 5 healthy adult participants received a single IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1 (Vaccination 1), 6 months (Booster 1) and 12 months (Booster 2). As per protocol amendment 10, after unblinding, enrolled participants who had initially received placebo were offered a single dose of 5*10^10 vp Ad26.COV2.S.
- COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10): Group 1 and 4 healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2) and matching placebo at 6 and 12 months after vaccination 2 as Booster 1 and Booster 2 vaccines. As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad hoc booster dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
- COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL: Group 2 healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1), Day 57 (Vaccination 2) and 6 months after Vaccination 2(Booster 1). At 12 months after vaccination 2, participants received placebo matching to Ad26.COV2.S vaccine (Booster 2).
- COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10: Group 3 healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2) and matching placebo at 6 months after vaccination 2 as Booster 1 vaccination and Ad26.COV2.S 5*10^10 vp at 12 months after vaccination 2 as Booster 2 vaccination.
- COHORT 2B: Placebo, B: PL: Group 5 healthy adult participants aged >=18 to <=55 received a single IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1 (Vaccination 1), Day 57 (Vaccination 2), 8 Month (Booster 1) and 14 months (Booster 2). As per protocol amendment 10, after unblinding, enrolled participants who had initially received placebo were offered a single dose of 5*10^10 vp Ad26.COV2.S.
- COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10): Adult participants (with good or stable health) aged >=65 years received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad hoc booster dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
- COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10): Adult participants (with good or stable health) aged >=65 years received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and matching placebo on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad hoc booster dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
- COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10): Adult participants (with good or stable health) aged >=65 years received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad hoc booster dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
- COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10): Adult participants (with good or stable health) aged >=65 years received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and matching placebo on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad hoc booster dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
- COHORT 3: Placebo, Placebo: Adult participants (with good or stable health) aged >=65 years received a single IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1 (vaccination1) and 57 (Vaccination2). As per protocol amendment 10, after unblinding, enrolled participants who had initially received placebo were offered a single dose of 5*10^10 vp Ad26.COV2.S.
Period: Overall Study
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Started | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5 | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15 | 81 | 80 | 82 | 79 | 81
Dose 1 | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5 | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15 | 81 | 80 | 82 | 79 | 81
Dose 2 | 74 | 74 | 74 | 67 | 74 | 4 | 5 | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 56 | 29 | 27 | 14 | 77 | 80 | 80 | 78 | 79
Ad Hoc Booster Dose | 6 | 8 | 7 | 7 | 0 | 1 | 2 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 7 | 0 | 0 | 0 | 11 | 15 | 14 | 9 | 0
Post Booster 1 Dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 42 | 19 | 20 | 1 | 45 | 21 | 20 | 0 | 0 | 0 | 0 | 0 | 0
Post Booster 2 Dose | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 13 | 10 | 0 | 8 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 48 | 49 | 42 | 39 | 36 | 3 | 5 | 4 | 4 | 4 | 33 | 15 | 14 | 7 | 31 | 16 | 15 | 5 | 65 | 53 | 53 | 57 | 6
Not Completed | 29 | 26 | 33 | 34 | 41 | 2 | 0 | 1 | 1 | 1 | 25 | 14 | 18 | 10 | 31 | 14 | 13 | 10 | 16 | 27 | 29 | 22 | 75
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 2 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 5 | 5 | 4 | 1 | 7 | 7 | 1 | 0 | 1 | 1 | 2 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 22 | 24 | 23 | 14 | 0 | 0 | 1 | 0 | 1 | 17 | 7 | 10 | 6 | 20 | 6 | 11 | 4 | 14 | 24 | 24 | 16 | 14
Not completed — Other | 3 | 2 | 5 | 9 | 23 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 2 | 3 | 0 | 0 | 6 | 1 | 0 | 2 | 2 | 60

BASELINE CHARACTERISTICS:
Groups:
- COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 5*10^10 vp on Day 1 (Vaccination 1) and matching placebo on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad AHBV of Ad26.COV2.S at the dose of 5*10^10 vp >=6 months after Vaccination 2.
- Total: Total of all reporting groups
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo | Total
Number analyzed (Participants) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5 | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15 | 81 | 80 | 82 | 79 | 81 | 1076
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.11) | 35.7 (9.99) | 34.5 (10.59) | 35.1 (10.48) | 35 (9.88) | 43 (11.45) | 44.4 (4.39) | 29.6 (4.34) | 41.2 (5.54) | 40.8 (11.97) | 36.8 (9.27) | 38.1 (9.98) | 39.2 (10.53) | 37.5 (10.41) | 37.6 (9.93) | 38.3 (9.81) | 36.1 (11.48) | 37 (9.99) | 69.5 (4.24) | 69.8 (3.74) | 69.7 (4.33) | 70.3 (4.18) | 69.9 (3.73) | 48.9 (18.27)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5 | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15 | 0 | 0 | 0 | 0 | 0 | 673
  From 65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 81 | 80 | 81 | 78 | 81 | 401
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 38 | 42 | 39 | 1 | 4 | 2 | 4 | 3 | 33 | 15 | 12 | 10 | 23 | 10 | 15 | 10 | 40 | 36 | 42 | 40 | 43 | 541
  Male | 36 | 37 | 37 | 31 | 38 | 4 | 1 | 3 | 1 | 2 | 25 | 14 | 20 | 7 | 39 | 20 | 13 | 5 | 41 | 44 | 40 | 39 | 38 | 535
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 2 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 4 | 2 | 5 | 2 | 2 | 3 | 0 | 1 | 2 | 0 | 3 | 46
  Not Hispanic or Latino | 73 | 69 | 73 | 71 | 72 | 5 | 5 | 4 | 5 | 4 | 55 | 26 | 28 | 14 | 56 | 28 | 25 | 12 | 81 | 78 | 80 | 79 | 78 | 1021
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
  Asian | 2 | 1 | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 2 | 1 | 2 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 4 | 3 | 9 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 2 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 38
  White | 71 | 71 | 70 | 66 | 65 | 4 | 4 | 4 | 5 | 5 | 49 | 22 | 28 | 15 | 55 | 22 | 26 | 14 | 80 | 77 | 80 | 78 | 81 | 992
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with solicited local AEs for 7 days after vaccination 1 in Cohorts 1a and 1b were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days post-vaccination 1 on Day 1 (Day 8)
Population: Full analysis set (FAS) included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5
Participants | 50 | 50 | 57 | 59 | 8 | 4 | 3 | 5 | 4 | 0

2. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with solicited local AEs for 7 days after vaccination 2 in Cohorts 1a and 1b were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after vaccination 2 on Day 57 (Day 64)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 74 | 74 | 74 | 67 | 74 | 4 | 5 | 5 | 5 | 5
Participants | 49 | 5 | 55 | 7 | 2 | 4 | 0 | 5 | 1 | 0

3. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited local AEs for 7 days after ad hoc booster vaccination in Cohorts 1a and 1b were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after ad hoc booster vaccination (Day 488 up to Day 604)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure. Here, 0 in the "Overall Number of Participants Analyzed" field signifies that no participants were available for the analysis because none of the participants received ad hoc booster vaccination in the respective arms.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 6 | 8 | 7 | 7 | 0 | 1 | 2 | 2 | 0 | 0
Participants | 5 | 5 | 6 | 5 |  | 0 | 1 | 2 |  |

4. Primary Outcome: Cohorts 2a and 2b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with solicited local AEs for 7 days after vaccination 1 in Cohorts 2a and 2b were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after Vaccination 1 on Day 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15
Participants | 48 | 24 | 19 | 4 | 52 | 23 | 18 | 0

5. Primary Outcome: Cohort 2a: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Booster Vaccination 1
Description: Number of participants with solicited local AEs for 7 days after booster vaccination 1 in Cohort 2a were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after booster vaccination 1 on Day 183 (Day 190)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 42 | 19 | 20 | 1
Participants | 6 | 15 | 3 | 0

6. Primary Outcome: Cohort 2a: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Booster Vaccination 2
Description: Number of participants with solicited local AEs for 7 days after booster vaccination 2 in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after booster vaccination 2 on Day 366 (Day 373)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure. Here, 0 in the "Overall Number of Participants Analyzed" field signifies that no participants were available for the analysis because none of the participants received booster vaccination 2 in the respective arm.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 19 | 13 | 10 | 0
Participants | 3 | 3 | 5 |

7. Primary Outcome: Cohort 2a: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited local AEs for 7 days after ad hoc booster vaccination in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after ad hoc booster vaccination (Day 384 up to Day 451)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who received Ad Hoc booster vaccination and were evaluable for this outcome measure. Here, 0 in the "Overall Number of Participants Analyzed" field signifies that no participants were available for the analysis because none of the participants received ad hoc booster vaccination in the respective arms.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 4 | 0 | 0 | 0
Participants | 1 |  |  |

8. Primary Outcome: Cohort 2b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with solicited local AEs for 7 days after Vaccination 2 in Cohort 2b were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after Vaccination 2 on Day 57 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 56 | 29 | 27 | 14
Participants | 42 | 21 | 18 | 3

9. Primary Outcome: Cohort 2b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Booster Vaccination 1
Description: Number of participants with solicited local AEs for 7 days after booster vaccination 1 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after booster vaccination 1 on Day 239 (Day 246)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure. Here, 0 in the "Overall Number of Participants Analyzed" field signifies that no participants were available for the analysis because none of the participants received booster vaccination 1 in the respective arm.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 45 | 21 | 20 | 0
Participants | 4 | 15 | 4 |

10. Primary Outcome: Cohort 2b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Booster Vaccination 2
Description: Number of participants with solicited local AEs for 7 days after booster Vaccination 2 in Cohort 2b were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after booster vaccination 2 on Day 422 (Day 429)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure. Here, 0 in the "Overall Number of Participants Analyzed" field signifies that no participants were available for the analysis because none of the participants received booster vaccination 2 in the respective arms.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 8 | 3 | 5 | 0
Participants | 0 | 1 | 4 |

11. Primary Outcome: Cohort 2b: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited local AEs for 7 days after ad hoc booster vaccination in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site).
Time Frame: 7 days after ad hoc booster vaccination (Day 369 up to Day 412)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants | 4 |  |  |

12. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with solicited systemic AEs for 7 days after vaccination 1 in Cohorts 1a and 1b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after vaccination 1 on Day 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5
Participants | 48 | 52 | 63 | 62 | 17 | 4 | 3 | 5 | 5 | 4

13. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with solicited systemic AEs for 7 days after vaccination 2 in Cohorts 1a and 1b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after Vaccination 2 on Day 57 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 74 | 74 | 74 | 67 | 74 | 4 | 5 | 5 | 5 | 5
Participants | 43 | 23 | 51 | 19 | 15 | 3 | 2 | 4 | 1 | 3

14. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited systemic AEs for 7 days after ad hoc booster vaccination in Cohorts 1a and 1b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post Ad Hoc Booster Vaccination (day of Ad hoc booster vaccination and the subsequent 7 days).
Time Frame: 7 days after ad hoc booster vaccination (Day 488 up to Day 604)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 6 | 8 | 7 | 7 | 0 | 1 | 2 | 2 | 0 | 0
Participants | 5 | 6 | 3 | 4 |  | 0 | 2 | 2 |  |

15. Primary Outcome: Cohorts 2a and 2b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with solicited systemic AEs for 7 days after vaccination 1 in Cohorts 2a and 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after Vaccination 1 on Day 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15
Participants | 47 | 23 | 21 | 8 | 50 | 23 | 21 | 5

16. Primary Outcome: Cohort 2a: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Booster Vaccination 1
Description: Number of participants with solicited systemic AEs for 7 days post booster vaccination 1 in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after booster vaccination 1 on Day 183 (Day 190)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 42 | 19 | 20 | 1
Participants | 14 | 11 | 5 | 0

17. Primary Outcome: Cohort 2a: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Booster Vaccination 2
Description: Number of participants with solicited systemic AEs for 7 days after booster vaccination 2 in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after booster vaccination 2 on Day 366 (Day 373)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 19 | 13 | 10 | 0
Participants | 6 | 2 | 2 |

18. Primary Outcome: Cohort 2a: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited systemic AEs for 7 days after ad hoc booster vaccination in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post adhoc booster vaccination (day of ad hoc booster vaccination and the subsequent 7 days).
Time Frame: 7 days after ad hoc booster vaccination (Day 384 up to Day 451)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 4 | 0 | 0 | 0
Participants | 1 |  |  |

19. Primary Outcome: Cohort 2b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with solicited systemic AEs for 7 days after vaccination 2 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after Vaccination 2 on Day 57 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 56 | 29 | 27 | 14
Participants | 40 | 17 | 15 | 6

20. Primary Outcome: Cohort 2b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Booster Vaccination 1
Description: Number of participants with solicited systemic AEs for 7 days after booster vaccination 1 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after booster vaccination 1 on Day 239 (Day 246)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 45 | 21 | 20 | 0
Participants | 14 | 13 | 4 |

21. Primary Outcome: Cohort 2b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Booster Vaccination 2
Description: Number of participants with solicited systemic AEs for 7 days after booster vaccination 2 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days after booster vaccination 2 on Day 422 (Day 429)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 8 | 3 | 5 | 0
Participants | 2 | 2 | 4 |

22. Primary Outcome: Cohort 2b: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited systemic AEs for 7 days after ad hoc booster vaccination in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post ad hoc booster vaccination (day of ad hoc booster vaccination and the subsequent 7 days).
Time Frame: 7 days after ad hoc booster vaccination (Day 369 up to Day 412)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants | 2 |  |  |

23. Primary Outcome: Cohort 3: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with solicited local AEs for 7 days after vaccination 1 in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site).
Time Frame: 7 days after vaccination 1 on Day 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 81 | 80 | 82 | 79 | 81
Participants | 38 | 30 | 33 | 34 | 7

24. Primary Outcome: Cohort 3: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with solicited systemic AEs for 7 days after vaccination 1 in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 1 on Day 1 (Day 8)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 81 | 80 | 82 | 79 | 81
Participants | 39 | 35 | 47 | 42 | 20

25. Primary Outcome: Cohort 3: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with solicited local AEs for 7 days after vaccination 2 in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site).
Time Frame: 7 days post-vaccination 2 on Day 57 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 77 | 80 | 80 | 78 | 79
Participants | 41 | 5 | 51 | 13 | 11

26. Primary Outcome: Cohort 3: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with solicited systemic AEs for 7 days after vaccination 2 in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 after post-vaccination 2 on Day 57 (Day 64)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 77 | 80 | 80 | 78 | 79
Participants | 33 | 24 | 40 | 24 | 24

27. Primary Outcome: Cohort 3: Number of Participants With Solicited Local (Injection Site) Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited local AEs for 7 days after ad hoc booster vaccination in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site).
Time Frame: 7 days after ad hoc booster vaccination (Day 456 up to Day 711)
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who received Ad Hoc booster vaccination and were evaluable for this outcome measure. Here, 0 in the "Overall Number of Participants Analyzed" field signifies that no participants were available for the analysis because none of the participants received ad hoc booster vaccination in the respective arm.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 11 | 15 | 14 | 9 | 0
Participants | 5 | 6 | 4 | 5 |

28. Primary Outcome: Cohort 3: Number of Participants With Solicited Systemic Adverse Events (AEs) for 7 Days After Ad Hoc Booster Vaccination
Description: Number of participants with solicited systemic AEs for 7 days after ad hoc booster vaccination in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post ad hoc booster vaccination (day of ad hoc booster vaccination and the subsequent 7 days).
Time Frame: 7 days after ad hoc booster vaccination (Day 456 up to Day 711)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 11 | 15 | 14 | 9 | 0
Participants | 3 | 7 | 4 | 6 |

29. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with unsolicited AEs after vaccination 1 in Cohorts 1a and 1b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after vaccination 1 on Day 1 (Day 29)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5
Participants | 11 | 20 | 26 | 24 | 14 | 2 | 3 | 4 | 4 | 2

30. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with unsolicited AEs after vaccination 2 in Cohorts 1a and 1b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after vaccination 2 on Day 57 (Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- COHORT 1A: Ad26 1e11, PL(,AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and matching placebo on Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single AHBV of Ad26.COV2.S at the dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(,AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 74 | 74 | 74 | 67 | 74 | 4 | 5 | 5 | 5 | 5
Participants | 10 | 4 | 7 | 12 | 6 | 2 | 0 | 1 | 0 | 1

31. Primary Outcome: Cohorts 1a and 1b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Ad Hoc Booster Vaccination
Description: Number of participants with unsolicited AEs after ad hoc booster vaccination in Cohorts 1a and 1b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after ad hoc booster vaccination (Day 488 up to Day 625)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 6 | 8 | 7 | 7 | 0 | 1 | 2 | 2 | 0 | 0
Participants | 0 | 1 | 1 | 0 |  | 0 | 0 | 0 |  |

32. Primary Outcome: Cohorts 2a and 2b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with unsolicited AEs after vaccination 1 in Cohorts 2a and 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after Vaccination 1 on Day 1 (Day 29)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15
Participants | 15 | 5 | 7 | 5 | 11 | 6 | 5 | 2

33. Primary Outcome: Cohort 2a: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Booster Vaccination 1
Description: Number of participants with unsolicited AEs after booster 1 vaccination in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after booster vaccination 1 on Day 183 (Day 211)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 42 | 19 | 20 | 1
Participants | 2 | 2 | 0 | 0

34. Primary Outcome: Cohort 2a: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Booster Vaccination 2
Description: Number of participants with unsolicited AEs after booster vaccination 2 in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after booster vaccination 2 on Day 366 (Day 394)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 19 | 13 | 10 | 0
Participants | 2 | 1 | 1 |

35. Primary Outcome: Cohort 2a: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Ad Hoc Booster Vaccination
Description: Number of participants with unsolicited AEs after ad hoc booster vaccination in Cohort 2a were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after ad hoc booster vaccination (Day 384 up to Day 472)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 4 | 0 | 0 | 0
Participants | 0 |  |  |

36. Primary Outcome: Cohort 2b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with unsolicited AEs after vaccination 1 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after Vaccination 2 on Day 57 (Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 56 | 29 | 27 | 14
Participants | 7 | 4 | 3 | 2

37. Primary Outcome: Cohort 2b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Booster Vaccination 1
Description: Number of participants with unsolicited AEs 28 days after booster vaccination 1 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after booster vaccination 1 on Day 239 (Day 267)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 45 | 21 | 20 | 0
Participants | 1 | 4 | 2 |

38. Primary Outcome: Cohort 2b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Booster Vaccination 2
Description: Number of participants with unsolicited AEs 28 days after booster vaccination 2 in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after booster vaccination 2 on Day 422 (Day 450)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 8 | 3 | 5 | 0
Participants | 0 | 0 | 0 |

39. Primary Outcome: Cohort 2b: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Ad Hoc Booster Vaccination
Description: Number of participants with unsolicited AEs 28 days after ad hoc booster vaccination in Cohort 2b were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after ad hoc booster vaccination (Day 369 up to Day 433)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 7 | 0 | 0 | 0
Participants | 0 |  |  |

40. Primary Outcome: Cohort 3: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Vaccination 1 in the Primary Regimen
Description: Number of participants with unsolicited AEs 28 days after vaccination 1 in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after vaccination 1 on Day 1 (Day 29)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 81 | 80 | 82 | 79 | 81
Participants | 16 | 13 | 19 | 26 | 16

41. Primary Outcome: Cohort 3: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Vaccination 2 in the Primary Regimen
Description: Number of participants with unsolicited AEs 28 days after vaccination 2 in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after vaccination 2 on Day 57 (Day 85)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 77 | 80 | 80 | 78 | 79
Participants | 11 | 9 | 12 | 12 | 9

42. Primary Outcome: Cohort 3: Number of Participants With Unsolicited Adverse Events (AEs) for 28 Days After Ad Hoc Booster Vaccination
Description: Number of participants with unsolicited AEs 28 days after ad hoc booster vaccination in Cohort 3 were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days after ad hoc booster vaccination (Day 456 up to Day 732)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 11 | 15 | 14 | 9 | 0
Participants | 1 | 0 | 3 | 1 |

43. Primary Outcome: Cohorts 1a and 1b and Cohort 3: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Time Frame: Day 1 up to 2 years after Vaccination 2 on Day 57 (Day 787)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5 | 81 | 80 | 82 | 79 | 81
Participants | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 2

44. Primary Outcome: Cohorts 2a and 2b: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 43
Time Frame: Day 1 up to 6 months post primary regimen (up to Day 183 for Cohort 2a; up to Day 239 for Cohort 2b)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15
Participants | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

45. Primary Outcome: Cohorts 1a, 1b and 3: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: Number of participants with AESIs was reported. AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Thrombosis with Thrombocytopenia Syndrome (TTS), a syndrome characterized by a combination of both a thrombotic event and thrombocytopenia, was considered to be an AESI in this study. A suspected TTS case was defined as: Thrombotic events: suspected deep vessel venous or arterial thrombotic events; Thrombocytopenia, defined as platelet count below 150,000/microliter.
Time Frame: Day 1 up to 2 years after Vaccination 2 on Day 57 (Day 787)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 77 | 75 | 75 | 73 | 77 | 5 | 5 | 5 | 5 | 5 | 81 | 80 | 82 | 79 | 81
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Primary Outcome: Cohorts 2a and 2b: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: as for outcome 45
Time Frame: Day 1 up to 6 months post primary regimen (up to Day 183 for Cohort 2a; up to Day 239 for Cohort 2b)
Population: FAS included all participants with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 58 | 29 | 32 | 17 | 62 | 30 | 28 | 15
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Cohort 1a: Percentage of Participants With Antibodies Binding to SARS-CoV-2 S Protein as Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Percentage of participants with antibodies binding to SARS-CoV-2 S protein as measured by ELISA was reported.
Time Frame: Days 29, 57, 71, 85, 239, and 422
Population: Per protocol immunogenicity (PPI) population included all randomized and vaccinated participants for whom immunogenicity data were available excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo
Number analyzed (Participants) | 65 | 64 | 67 | 64 | 70
Percentage of participants
  Day 29: number analyzed (Participants) | 64 | 63 | 67 | 64 | 70
  Day 29 | 98.4 [91.5 to 100.0] | 98.4 [91.5 to 100.0] | 100.0 [94.6 to 100.0] | 98.4 [91.6 to 100.0] | 1.4 [0.0 to 7.7]
  Day 57: number analyzed (Participants) | 65 | 64 | 66 | 61 | 66
  Day 57 | 100.0 [94.4 to 100.0] | 98.4 [91.6 to 100.0] | 100.0 [94.6 to 100.0] | 96.7 [88.7 to 99.6] | 1.5 [0.0 to 8.2]
  Day 71: number analyzed (Participants) | 62 | 59 | 64 | 56 | 61
  Day 71 | 100.0 [94.1 to 100.0] | 100.0 [93.9 to 100.0] | 100.0 [94.4 to 100.0] | 96.4 [87.7 to 99.6] | 1.6 [0.0 to 8.8]
  Day 85: number analyzed (Participants) | 65 | 61 | 63 | 58 | 64
  Day 85 | 100.0 [94.3 to 100.0] | 98.4 [91.2 to 100.0] | 100.0 [94.3 to 100.0] | 96.6 [88.1 to 99.6] | 4.7 [1.0 to 13.1]
  Day 239: number analyzed (Participants) | 61 | 59 | 56 | 52 | 49
  Day 239 | 100.0 [94.0 to 100.0] | 98.3 [90.9 to 100.0] | 100.0 [93.6 to 100.0] | 94.2 [84.1 to 98.8] | 2.0 [0.1 to 10.9]
  Day 422: number analyzed (Participants) | 44 | 50 | 46 | 42 | 6
  Day 422 | 100.0 [91.8 to 100.0] | 92.0 [80.8 to 97.8] | 100.0 [92.3 to 100.0] | 100.0 [91.6 to 100.0] | 66.7 [22.3 to 95.7]

48. Secondary Outcome: Cohort 1b: Percentage of Participants With Antibodies Binding to SARS-CoV-2 S Protein as Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Percentage of participants with antibodies binding to SARS-CoV-2 S protein as measured by ELISA was reported.
Time Frame: Days 29 and 71
Population: PPI population included all randomized and vaccinated participants for whom immunogenicity data were available excluding participants with major protocol deviations expecting to impact the immunogenicity outcomes. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 4
Percentage of participants
  Day 29 | 80.0 [28.4 to 99.5] | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 0.0 [0.0 to 60.2]
  Day 71: number analyzed (Participants) | 4 | 5 | 5 | 5 | 4
  Day 71 | 100.0 [39.8 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 100.0 [47.8 to 100.0] | 0.0 [0.0 to 60.2]

49. Secondary Outcome: Cohorts 2a: Percentage of Participants With Antibodies Binding to SARS-CoV-2 S Protein as Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Percentage of participants with antibodies binding to SARS-CoV-2 S protein as measured by ELISA was reported.
Time Frame: Days 8, 29, 183, 190, 211, 366, 373, and 394,
Population: PPI population was analyzed. Here, 'N' (Overall number of participants analyzed) =participants who were evaluable for this outcome measure and "n" (number analyzed) =participants who were evaluable for specified time points. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 51 | 23 | 26 | 15
Percentage of participants
  Day 8: number analyzed (Participants) | 50 | 23 | 26 | 15
  Day 8 | 6.0 [1.3 to 16.5] | 0.0 [0.0 to 14.8] | 0.0 [0.0 to 13.2] | 0.0 [0.0 to 21.8]
  Day 29 | 98.0 [89.4 to 99.9] | 100.0 [85.2 to 100.0] | 100.0 [86.8 to 100.0] | 6.7 [0.2 to 31.9]
  Day 183: number analyzed (Participants) | 34 | 18 | 15 | 1
  Day 183 | 97.0 [84.2 to 99.9] | 100.0 [81.5 to 100.0] | 86.7 [59.5 to 98.3] | 100.0 [2.5 to 100.0]
  Day 190: number analyzed (Participants) | 32 | 16 | 13 | 1
  Day 190 | 96.8 [83.3 to 99.9] | 100.0 [79.4 to 100.0] | 92.3 [64.0 to 99.8] | 100.0 [2.5 to 100.0]
  Day 211: number analyzed (Participants) | 28 | 14 | 14 | 1
  Day 211 | 100.0 [87.2 to 100.0] | 100.0 [76.8 to 100.0] | 85.7 [57.2 to 98.2] | 100.0 [2.5 to 100.0]
  Day 366: number analyzed (Participants) | 21 | 13 | 6 | 0
  Day 366 | 95.2 [76.2 to 99.9] | 100.0 [75.3 to 100.0] | 83.3 [35.9 to 99.6] |
  Day 373: number analyzed (Participants) | 17 | 11 | 4 | 0
  Day 373 | 94.1 [71.3 to 99.9] | 100.0 [71.5 to 100.0] | 100.0 [39.8 to 100.0] |
  Day 394: number analyzed (Participants) | 13 | 11 | 3 | 0
  Day 394 | 92.3 [64.0 to 99.8] | 100.0 [71.5 to 100.0] | 100.0 [29.2 to 100.0] |

50. Secondary Outcome: Cohort 2b: Percentage of Participants With Antibodies Binding to SARS-CoV-2 S Protein as Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Percentage of participants with antibodies binding to SARS-CoV-2 S protein as measured by ELISA was reported.
Time Frame: Days 8, 29, 57, 64, 85, 239, 246, 267 and 422
Population: PPI population was analyzed. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 51 | 28 | 24 | 12
Percentage of participants
  Day 8: number analyzed (Participants) | 51 | 26 | 23 | 12
  Day 8 | 0.0 [0.0 to 7.0] | 3.8 [0.1 to 19.6] | 4.5 [0.1 to 22.8] | 0.0 [0.0 to 26.5]
  Day 29: number analyzed (Participants) | 49 | 28 | 24 | 12
  Day 29 | 95.9 [86.0 to 99.5] | 96.4 [81.7 to 99.9] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 26.5]
  Day 57: number analyzed (Participants) | 49 | 26 | 24 | 12
  Day 57 | 95.8 [85.7 to 99.5] | 100.0 [86.8 to 100.0] | 100.0 [84.6 to 100.0] | 0.0 [0.0 to 26.5]
  Day 64: number analyzed (Participants) | 46 | 24 | 23 | 11
  Day 64 | 100.0 [92.1 to 100.0] | 100.0 [85.8 to 100.0] | 100.0 [83.9 to 100.0] | 0.0 [0.0 to 28.5]
  Day 85: number analyzed (Participants) | 46 | 26 | 21 | 11
  Day 85 | 97.8 [88.2 to 99.9] | 100.0 [86.8 to 100.0] | 100.0 [82.4 to 100.0] | 0.0 [0.0 to 28.5]
  Day 239: number analyzed (Participants) | 40 | 22 | 20 | 0
  Day 239 | 97.4 [86.5 to 99.9] | 95.5 [77.2 to 99.9] | 94.4 [72.7 to 99.9] |
  Day 246: number analyzed (Participants) | 38 | 15 | 17 | 0
  Day 246 | 97.4 [86.2 to 99.9] | 100.0 [78.2 to 100.0] | 93.8 [69.8 to 99.8] |
  Day 267: number analyzed (Participants) | 37 | 18 | 18 | 0
  Day 267 | 97.2 [85.5 to 99.9] | 100.0 [81.5 to 100.0] | 93.8 [69.8 to 99.8] |
  Day 422: number analyzed (Participants) | 5 | 3 | 4 | 0
  Day 422 | 100.0 [47.8 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] |

51. Secondary Outcome: Cohort 3: Percentage of Participants With Antibodies Binding to SARS-CoV-2 S Protein as Measured by Enzyme-linked Immunosorbent Assay (ELISA)
Description: Percentage of participants with antibodies binding to SARS-CoV-2 S protein as measured by ELISA was reported.
Time Frame: Days 15, 29, 87, 100, 114 and 268
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 72 | 73 | 74 | 75 | 75
Percentage of participants
  Day 15: number analyzed (Participants) | 59 | 58 | 55 | 62 | 61
  Day 15 | 78.0 [65.3 to 87.7] | 72.4 [59.1 to 83.3] | 79.6 [66.5 to 89.4] | 77.4 [65.0 to 87.1] | 1.6 [0.0 to 8.8]
  Day 29 | 95.8 [88.3 to 99.1] | 97.2 [90.3 to 99.7] | 95.8 [88.3 to 99.1] | 97.3 [97.3 to 99.7] | 0.0 [0.0 to 4.9]
  Day 87: number analyzed (Participants) | 67 | 67 | 66 | 71 | 69
  Day 87 | 97.0 [89.6 to 99.6] | 97.0 [89.5 to 99.6] | 96.9 [89.2 to 99.6] | 98.6 [92.4 to 100.0] | 1.5 [0.0 to 7.9]
  Day 100: number analyzed (Participants) | 64 | 69 | 66 | 70 | 68
  Day 100 | 98.4 [91.6 to 100.0] | 97.1 [89.8 to 99.6] | 98.4 [91.6 to 100.0] | 98.6 [92.3 to 100.0] | 0.0 [0.0 to 5.4]
  Day 114: number analyzed (Participants) | 66 | 68 | 66 | 71 | 69
  Day 114 | 98.5 [91.8 to 100.0] | 97.0 [89.6 to 99.6] | 98.4 [91.6 to 100.0] | 98.6 [92.4 to 100.0] | 1.5 [0.0 to 7.9]
  Day 268: number analyzed (Participants) | 60 | 56 | 55 | 57 | 6
  Day 268 | 98.3 [91.1 to 100.0] | 85.5 [73.3 to 93.5] | 100.0 [93.3 to 100.0] | 87.7 [76.3 to 94.9] | 16.7 [0.4 to 64.1]

52. Secondary Outcome: Cohort 1a: Geometric Mean Titers (GMTs) of SARS-CoV-2 Neutralizing Antibodies to the Wild Type Virus as Measured by Virus Neutralization Assay (VNA)
Description: GMTs of SARS-CoV-2 neutralizing antibodies to the Wild-type VNA were reported.
Time Frame: Days 29, 57, 71, 85, 239 and 422
Population: PPI population was analyzed. 'N' (Overall number of participants analyzed) =participants who were evaluable for this outcome measure and "n" (number analyzed) =participants who were evaluable for specified time points. Due to the change in planned analysis, data was not collected and analyzed for Cohort 1b and thus no data was reported for this outcome measure. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo
Number analyzed (Participants) | 22 | 24 | 24 | 23 | 25
Titers
  Day 29 | 233 [170 to 319] | 224 [158 to 319] | 333 [206 to 537] | 219 [170 to 282] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 57: number analyzed (Participants) | 22 | 24 | 22 | 21 | 23
  Day 57 | 310 [232 to 414] | 284 [220 to 367] | 458 [309 to 677] | 392 [273 to 563] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 71: number analyzed (Participants) | 21 | 23 | 23 | 20 | 22
  Day 71 | 862 [666 to 1115] | 294 [229 to 378] | 1189 [845 to 1672] | 414 [310 to 553] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 85: number analyzed (Participants) | 21 | 23 | 23 | 20 | 22
  Day 85 | 919 [727 to 1161] | 317 [217 to 463] | 1127 [801 to 1587] | 422 [305 to 584] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (61).
  Day 239: number analyzed (Participants) | 21 | 21 | 20 | 20 | 19
  Day 239 | 465 [338 to 641] | 215 [146 to 317] | 771 [514 to 1154] | 408 [232 to 716] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 422: number analyzed (Participants) | 17 | 19 | 19 | 18 | 0
  Day 422 | 328 [202 to 531] | 235 [132 to 418] | 425 [294 to 613] | 307 [205 to 460] |

53. Secondary Outcome: Cohorts 2a: Geometric Mean Titers (GMTs) of SARS-CoV-2 Neutralizing Antibodies to the Wild Type Virus as Measured by Virus Neutralization Assay (VNA)
Description: GMTs of SARS-CoV-2 neutralizing antibodies to the Wild-type VNA were reported.
Time Frame: Days 29, 183, 190, 211, 366, 373 and 394
Population: PPI population was analyzed. Here, 'N' (Overall number of participants analyzed) =participants who were evaluable for this outcome measure and "n" (number analyzed) =participants who were evaluable for specified time points. Due to the change in planned analysis, data was not collected and analyzed for Cohort 2b and thus no data was reported for this outcome measure. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 51 | 23 | 26 | 15
Titers
  Day 29 | 311 [235 to 411] | 326 [258 to 411] | 369 [251 to 542] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 183: number analyzed (Participants) | 34 | 18 | 15 | 1
  Day 183 | 241 [179 to 324] | 379 [214 to 672] | 172 [107 to 277] | 833 [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 190: number analyzed (Participants) | 32 | 16 | 13 | 1
  Day 190 | 208 [149 to 290] | 1576 [976 to 2544] | 162 [88 to 301] | 961 [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 211: number analyzed (Participants) | 28 | 14 | 14 | 1
  Day 211 | 216 [150 to 311] | 2035 [1202 to 3446] | 157 [96 to 256] | 486 [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 366: number analyzed (Participants) | 21 | 13 | 6 | 0
  Day 366 | 224 [131 to 383] | 1137 [661 to 1955] | 124 [60 to 258] |
  Day 373: number analyzed (Participants) | 17 | 11 | 4 | 0
  Day 373 | 245 [138 to 435] | 1248 [566 to 2753] | 973 [240 to 3954] |
  Day 394: number analyzed (Participants) | 13 | 11 | 3 | 0
  Day 394 | 297 [152 to 581] | 1387 [612 to 3143] | 3061 [141 to NA] — Upper limit of 95% CI could not be estimated as the value was above the upper limit of quantification (ULOQ) (12800). |

54. Secondary Outcome: Cohort 3: Geometric Mean Titers (GMTs) of SARS-CoV-2 Neutralizing Antibodies to the Wild Type Virus as Measured by Virus Neutralization Assay (VNA)
Description: GMTs of SARS-CoV-2 neutralizing antibodies to the Wild-type VNA were reported.
Time Frame: Days 15, 29, 87, 100, 114 and 268
Population: FAS included all participants with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 23 | 24 | 25 | 23 | 22
Titers
  Day 15: number analyzed (Participants) | 11 | 10 | 14 | 10 | 10
  Day 15 | 190 [100 to 360] | 153 [90 to 261] | 209 [121 to 361] | 140 [70 to 280] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 29 | 267 [183 to 389] | 229 [152 to 346] | 261 [168 to 406] | 174 [131 to 233] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 87: number analyzed (Participants) | 19 | 21 | 22 | 20 | 19
  Day 87 | 224 [134 to 375] | 165 [114 to 238] | 245 [174 to 346] | 198 [126 to 309] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 100: number analyzed (Participants) | 19 | 22 | 22 | 19 | 19
  Day 100 | 878 [521 to 1478] | 168 [106 to 266] | 574 [367 to 897] | 178 [97 to 329] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 114: number analyzed (Participants) | 19 | 22 | 22 | 19 | 19
  Day 114 | 954 [551 to 1652] | 164 [98 to 273] | 895 [498 to 1609] | 158 [78 to 319] | NA [NA to NA] — Data could not be estimated as the value was below the LLOQ (58).
  Day 268: number analyzed (Participants) | 0 | 19 | 0 | 0 | 0
  Day 268 |  | 114 [65 to 201] |  |  |

55. Secondary Outcome: Cohort 1a: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: Interferon Gamma (IFNg)+ or Interleukin 2+ (IL2+) Not Helper Cell Type 2 (TH2)
Description: Percentage of participants with SARS-Cov2 S Specific CD4+ T-cell Responses for IFNg+ or IL2+ not Helper cell type 2 (TH2) was reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination.
Time Frame: Baseline, Days 15, 29, 57, 71, 85, 239 and 422
Population: PPI population was analyzed. Here, 'N' (Overall number of participants analyzed) =participants who were evaluable for this outcome measure and "n" (number analyzed) =participants who were evaluable for specified time points. Due to the change in planned analysis, data was not collected and analyzed for Cohort 1b and thus no data was reported for this outcome measure. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo
Number analyzed (Participants) | 37 | 39 | 36 | 35 | 39
Percentage of participants
  Baseline: number analyzed (Participants) | 37 | 39 | 35 | 35 | 39
  Baseline | 8 [2 to 22] | 8 [2 to 21] | 0 [0 to 10] | 3 [0 to 15] | 0 [0 to 9]
  Day 15: number analyzed (Participants) | 37 | 38 | 36 | 34 | 39
  Day 15 | 76 [59 to 88] | 76 [60 to 89] | 83 [67 to 94] | 82 [65 to 93] | 8 [2 to 21]
  Day 29: number analyzed (Participants) | 37 | 37 | 36 | 32 | 37
  Day 29 | 73 [56 to 86] | 70 [53 to 84] | 78 [61 to 90] | 72 [53 to 86] | 19 [8 to 35]
  Day 57: number analyzed (Participants) | 36 | 36 | 35 | 30 | 33
  Day 57 | 75 [58 to 88] | 53 [35 to 70] | 77 [60 to 90] | 63 [44 to 80] | 12 [3 to 28]
  Day 71: number analyzed (Participants) | 35 | 36 | 34 | 28 | 32
  Day 71 | 63 [45 to 79] | 47 [30 to 65] | 91 [76 to 98] | 61 [41 to 79] | 16 [5 to 33]
  Day 85: number analyzed (Participants) | 37 | 35 | 33 | 29 | 34
  Day 85 | 68 [50 to 82] | 46 [29 to 63] | 85 [68 to 95] | 59 [39 to 76] | 12 [3 to 27]
  Day 239: number analyzed (Participants) | 34 | 34 | 12 | 13 | 0
  Day 239 | 47 [30 to 65] | 47 [30 to 65] | 75 [43 to 95] | 38 [14 to 68] |
  Day 422: number analyzed (Participants) | 22 | 23 | 13 | 11 | 0
  Day 422 | 27 [11 to 50] | 43 [23 to 66] | 54 [25 to 81] | 36 [11 to 69] |

56. Secondary Outcome: Cohorts 2a: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: Interferon Gamma (IFNg)+ or Interleukin 2+ (IL2+) Not Helper Cell Type 2 (TH2)
Description: as for outcome 55
Time Frame: Baseline, Days 29 and 366
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 11 | 5 | 5 | 3
Percentage of participants
  Baseline | 9 [0 to 41] | 20 [1 to 72] | 0 [0 to 52] | 33 [1 to 91]
  Day 29 | 82 [48 to 98] | 100 [48 to 100.0] | 80 [28 to 99] | 0 [0 to 71]
  Day 366: number analyzed (Participants) | 9 | 5 | 3 | 0
  Day 366 | 11 [0 to 48] | 20 [1 to 72] | 0 [0 to 71] |

57. Secondary Outcome: Cohort 2b: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: Interferon Gamma (IFNg)+ or Interleukin 2+ (IL2+) Not Helper Cell Type 2 (TH2)
Description: as for outcome 55
Time Frame: Baseline, Days 29, 57, 85 and 422
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 12 | 5 | 6 | 2
Percentage of participants
  Baseline | 25 [5 to 57] | 20 [1 to 72] | 17 [0 to 64] | 0 [0 to 84]
  Day 29: number analyzed (Participants) | 11 | 5 | 6 | 2
  Day 29 | 82 [48 to 98] | 40 [5 to 85] | 67 [22 to 96] | 0 [0 to 84]
  Day 57: number analyzed (Participants) | 12 | 5 | 5 | 2
  Day 57 | 75 [43 to 95] | 80 [28 to 99] | 40 [5 to 85] | 0 [0 to 84]
  Day 85: number analyzed (Participants) | 10 | 5 | 6 | 2
  Day 85 | 60 [26 to 88] | 80 [28 to 99] | 50 [12 to 88] | 0 [0 to 84]
  Day 422: number analyzed (Participants) | 1 | 1 | 1 | 0
  Day 422 | 0 [0 to 98] | 0 [0 to 98] | 100 [3 to 100] |

58. Secondary Outcome: Cohort 3: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: IFNg+ or IL2+ Not Helper Cell Type 2 (TH2)
Description: as for outcome 55
Time Frame: Baseline, Days 15, 29, 87, 100, 114 and 268
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 38 | 36 | 34 | 41 | 35
Percentage of participants
  Baseline: number analyzed (Participants) | 37 | 35 | 33 | 40 | 35
  Baseline | 0 [0 to 9] | 0 [0 to 10] | 3 [0 to 16] | 0 [0 to 9] | 6 [1 to 19]
  Day 15: number analyzed (Participants) | 38 | 35 | 33 | 39 | 35
  Day 15 | 61 [43 to 76] | 63 [45 to 79] | 67 [48 to 82] | 62 [45 to 77] | 6 [1 to 19]
  Day 29 | 66 [49 to 80] | 69 [52 to 84] | 68 [49 to 83] | 76 [60 to 88] | 14 [5 to 30]
  Day 87: number analyzed (Participants) | 31 | 27 | 23 | 33 | 26
  Day 87 | 42 [25 to 61] | 48 [29 to 68] | 39 [20 to 61] | 52 [34 to 69] | 4 [0 to 20]
  Day 100: number analyzed (Participants) | 33 | 33 | 27 | 36 | 30
  Day 100 | 61 [42 to 77] | 61 [42 to 77] | 78 [58 to 91] | 58 [41 to 74] | 3 [0 to 17]
  Day 114: number analyzed (Participants) | 34 | 32 | 29 | 36 | 29
  Day 114 | 71 [53 to 85] | 69 [50 to 84] | 69 [49 to 85] | 44 [28 to 62] | 17 [6 to 36]
  Day 268: number analyzed (Participants) | 29 | 26 | 10 | 14 | 0
  Day 268 | 59 [39 to 76] | 73 [52 to 88] | 40 [12 to 74] | 57 [29 to 82] |

59. Secondary Outcome: Cohort 1a: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: IL4+ and/or (IL5+/IL13+) and CD40L+
Description: Percentage of participants with SARS-Cov2 S Specific CD4+ T-cell responses for IL4+ and/or (IL5+/IL13+) and CD40L+ was reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination.
Time Frame: Baseline, Day 15, 29, 57, 71, 85, 239 and 422
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo
Number analyzed (Participants) | 37 | 39 | 36 | 35 | 39
Percentage of participants
  Baseline: number analyzed (Participants) | 37 | 39 | 35 | 35 | 39
  Baseline | 0 [0 to 9] | 0 [0 to 9] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 9]
  Day 15: number analyzed (Participants) | 37 | 38 | 36 | 34 | 39
  Day 15 | 0 [0 to 9] | 3 [0 to 14] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 9]
  Day 29: number analyzed (Participants) | 37 | 37 | 36 | 32 | 37
  Day 29 | 0 [0 to 9] | 0 [0 to 9] | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 9]
  Day 57: number analyzed (Participants) | 36 | 36 | 35 | 30 | 33
  Day 57 | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 12] | 6 [1 to 20]
  Day 71: number analyzed (Participants) | 35 | 36 | 34 | 28 | 32
  Day 71 | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 10] | 4 [0 to 18] | 0 [0 to 11]
  Day 85: number analyzed (Participants) | 37 | 35 | 33 | 29 | 34
  Day 85 | 0 [0 to 9] | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 12] | 0 [0 to 10]
  Day 239: number analyzed (Participants) | 34 | 34 | 12 | 13 | 0
  Day 239 | 3 [0 to 15] | 6 [1 to 20] | 17 [2 to 48] | 0 [0 to 25] |
  Day 422: number analyzed (Participants) | 22 | 23 | 13 | 11 | 0
  Day 422 | 5 [0 to 23] | 4 [0 to 22] | 0 [0 to 25] | 9 [0 to 41] |

60. Secondary Outcome: Cohort 2a: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: IL4+ and/or (IL5+/IL13+) and CD40L+
Description: as for outcome 59
Time Frame: Baseline, Days 29 and 366
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 11 | 5 | 5 | 3
Percentage of participants
  Baseline | 0 [0 to 28] | 0 [0 to 52] | 0 [0 to 52] | 0 [0 to 71]
  Day 29 | 0 [0 to 28] | 0 [0 to 52] | 0 [0 to 52] | 0 [0 to 71]
  Day 366: number analyzed (Participants) | 9 | 5 | 3 | 0
  Day 366 | 0 [0 to 34] | 0 [0 to 52] | 0 [0 to 71] |

61. Secondary Outcome: Cohort 2b: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: IL4+ and/or (IL5+/IL13+) and CD40L+
Description: as for outcome 59
Time Frame: Baseline, Days 29, 57, 85 and 422
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 12 | 5 | 6 | 2
Percentage of participants
  Baseline | 0 [0 to 26] | 0 [0 to 52] | 0 [0 to 46] | 0 [0 to 84]
  Day 29: number analyzed (Participants) | 11 | 5 | 6 | 2
  Day 29 | 0 [0 to 28] | 0 [0 to 52] | 0 [0 to 46] | 0 [0 to 84]
  Day 57: number analyzed (Participants) | 12 | 5 | 5 | 2
  Day 57 | 0 [0 to 26] | 0 [0 to 52] | 0 [0 to 52] | 0 [0 to 84]
  Day 85: number analyzed (Participants) | 10 | 5 | 6 | 2
  Day 85 | 0 [0 to 31] | 0 [0 to 52] | 0 [0 to 46] | 0 [0 to 84]
  Day 422: number analyzed (Participants) | 1 | 1 | 1 | 0
  Day 422 | 0 [0 to 98] | 0 [0 to 98] | 0 [0 to 98] |

62. Secondary Outcome: Cohort 3: Percentage of Participants With SARS-Cov2 S Specific CD4+ T-cell Responses: IL4+ and/or (IL5+/IL13+) and CD40L+
Description: as for outcome 59
Time Frame: Baseline, Days 15, 29, 87, 100, 114 and 268
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- COHORT 3: Placebo, PlaceboEdit Adult: Adult participants (with good or stable health) aged >=65 years received a single IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1 (vaccination1) and 57 (Vaccination2). As per protocol amendment 10, after unblinding, enrolled participants who had initially received placebo were offered a single dose of 5*10^10 vp Ad26.COV2.S.
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, PlaceboEdit Adult
Number analyzed (Participants) | 38 | 36 | 34 | 41 | 35
Percentage of participants
  Baseline: number analyzed (Participants) | 37 | 35 | 33 | 40 | 35
  Baseline | 0 [0 to 9] | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 9] | 0 [0 to 10]
  Day 15: number analyzed (Participants) | 38 | 35 | 33 | 39 | 35
  Day 15 | 0 [0 to 9] | 0 [0 to 10] | 3 [0 to 16] | 0 [0 to 9] | 0 [0 to 10]
  Day 29 | 0 [0 to 9] | 0 [0 to 10] | 0 [0 to 10] | 0 [0 to 9] | 0 [0 to 10]
  Day 87: number analyzed (Participants) | 31 | 27 | 23 | 33 | 26
  Day 87 | 0 [0 to 11] | 0 [0 to 13] | 4 [0 to 22] | 0 [0 to 11] | 0 [0 to 13]
  Day 100: number analyzed (Participants) | 33 | 33 | 27 | 36 | 30
  Day 100 | 6 [1 to 20] | 0 [0 to 11] | 0 [0 to 13] | 0 [0 to 10] | 0 [0 to 12]
  Day 114: number analyzed (Participants) | 34 | 32 | 29 | 36 | 29
  Day 114 | 0 [0 to 10] | 0 [0 to 11] | 0 [0 to 12] | 0 [0 to 10] | 0 [0 to 12]
  Day 268: number analyzed (Participants) | 29 | 26 | 10 | 14 | 0
  Day 268 | 7 [1 to 23] | 8 [1 to 25] | 20 [3 to 56] | 7 [0 to 34] |

63. Secondary Outcome: Cohort 1a: Percentage of Participants With SARS-Cov2 S Specific CD8+ T-cell Responses: IFNg+ or IL2+
Description: Percentage of participants with SARS-Cov2 S Specific CD8+ T-cell Responses for IFNg+ or IL2+ was reported. Cellular immunogenicity was measured by intracellular cytokine staining (ICS), allowing characterization of individual CD4 and CD8 T cell immune responses to vaccination.
Time Frame: Baseline, Days 15, 29, 57, 71, 85, 239 and 422
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo
Number analyzed (Participants) | 37 | 39 | 36 | 35 | 39
Percentage of participants
  Baseline: number analyzed (Participants) | 37 | 39 | 35 | 35 | 39
  Baseline | 0 [0 to 9] | 3 [0 to 13] | 0 [0 to 10] | 3 [0 to 15] | 5 [1 to 17]
  Day 15: number analyzed (Participants) | 37 | 38 | 36 | 34 | 39
  Day 15 | 54 [37 to 71] | 45 [29 to 62] | 56 [38 to 72] | 71 [53 to 85] | 8 [2 to 21]
  Day 29: number analyzed (Participants) | 37 | 37 | 36 | 32 | 37
  Day 29 | 68 [50 to 82] | 59 [42 to 75] | 81 [64 to 92] | 75 [57 to 89] | 3 [0 to 14]
  Day 57: number analyzed (Participants) | 36 | 36 | 35 | 30 | 33
  Day 57 | 72 [55 to 86] | 81 [64 to 92] | 89 [73 to 97] | 83 [65 to 94] | 6 [1 to 20]
  Day 71: number analyzed (Participants) | 34 | 36 | 35 | 28 | 32
  Day 71 | 68 [49 to 83] | 72 [55 to 86] | 86 [70 to 95] | 79 [59 to 92] | 9 [2 to 25]
  Day 85: number analyzed (Participants) | 37 | 35 | 33 | 29 | 34
  Day 85 | 73 [56 to 86] | 69 [51 to 83] | 88 [72 to 97] | 83 [64 to 94] | 9 [2 to 24]
  Day 239: number analyzed (Participants) | 34 | 34 | 12 | 13 | 0
  Day 239 | 62 [44 to 78] | 62 [44 to 78] | 92 [62 to 100] | 85 [55 to 98] |
  Day 422: number analyzed (Participants) | 23 | 23 | 13 | 11 | 0
  Day 422 | 52 [31 to 73] | 57 [34 to 77] | 77 [46 to 95] | 82 [48 to 98] |

64. Secondary Outcome: Cohort 2a: Percentage of Participants With SARS-Cov2 S Specific CD8+ T-cell Responses: IFNg+ or IL2+
Description: as for outcome 63
Time Frame: Baseline, Days 29 and 366
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 11 | 5 | 5 | 3
Percentage of participants
  Baseline | 0 [0 to 28] | 0 [0 to 52] | 0 [0 to 52] | 0 [0 to 71]
  Day 29 | 91 [59 to 100] | 100 [48 to 100] | 100 [48 to 100] | 0 [0 to 71]
  Day 366: number analyzed (Participants) | 9 | 4 | 3 | 0
  Day 366 | 78 [40 to 97] | 75 [19 to 99] | 100 [29 to 100] |

65. Secondary Outcome: Cohort 2b: Percentage of Participants With SARS-Cov2 S Specific CD8+ T-cell Responses: IFNg+ or IL2+
Description: as for outcome 63
Time Frame: Baseline, Days 29, 57, 85 and 422
Population: as for outcome 49
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 12 | 5 | 6 | 2
Percentage of participants
  Baseline | 8 [0 to 38] | 20 [1 to 72] | 0 [0 to 46] | 0 [0 to 84]
  Day 29: number analyzed (Participants) | 11 | 5 | 6 | 2
  Day 29 | 82 [48 to 98] | 80 [28 to 99] | 83 [36 to 100] | 0 [0 to 84]
  Day 57: number analyzed (Participants) | 12 | 5 | 5 | 2
  Day 57 | 92 [62 to 100] | 100 [48 to 100] | 80 [28 to 99] | 0 [0 to 84]
  Day 85: number analyzed (Participants) | 10 | 5 | 6 | 2
  Day 85 | 80 [44 to 97] | 100 [48 to 100] | 83 [36 to 100] | 0 [0 to 84]
  Day 422: number analyzed (Participants) | 1 | 1 | 1 | 0
  Day 422 | 100 [3 to 100] | 100 [3 to 100] | 100 [3 to 100] |

66. Secondary Outcome: Cohort 3: Percentage of Participants With SARS-Cov2 S Specific CD8+ T-cell Responses: IFNg+ or IL2+
Description: as for outcome 63
Time Frame: Baseline, Days 15, 29, 87, 100, 114 and 268
Population: as for outcome 54
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 36 | 35 | 33 | 39 | 33
Percentage of participants
  Baseline: number analyzed (Participants) | 36 | 34 | 31 | 39 | 31
  Baseline | 3 [0 to 15] | 0 [0 to 10] | 6 [1 to 21] | 0 [0 to 9] | 0 [0 to 11]
  Day 15: number analyzed (Participants) | 34 | 35 | 31 | 38 | 33
  Day 15 | 35 [20 to 54] | 23 [10 to 40] | 26 [12 to 45] | 26 [13 to 43] | 3 [0 to 16]
  Day 29 | 58 [41 to 74] | 51 [34 to 69] | 52 [34 to 69] | 64 [47 to 79] | 0 [0 to 11]
  Day 87: number analyzed (Participants) | 29 | 26 | 22 | 31 | 23
  Day 87 | 59 [39 to 76] | 58 [37 to 77] | 45 [24 to 68] | 71 [52 to 86] | 0 [0 to 15]
  Day 100: number analyzed (Participants) | 31 | 33 | 26 | 36 | 27
  Day 100 | 65 [45 to 81] | 52 [34 to 69] | 65 [44 to 83] | 67 [49 to 81] | 0 [0 to 13]
  Day 114: number analyzed (Participants) | 32 | 32 | 26 | 34 | 26
  Day 114 | 75 [57 to 89] | 47 [29 to 65] | 62 [41 to 80] | 68 [49 to 83] | 0 [0 to 13]
  Day 268: number analyzed (Participants) | 28 | 26 | 9 | 14 | 0
  Day 268 | 57 [37 to 76] | 50 [30 to 70] | 78 [40 to 97] | 71 [42 to 92] |

67. Secondary Outcome: Cohort 1a: Percentage of Participants With T Helper Cell 1/T Helper Cell 2 Ratio (Th1/Th2) Greater Than or Equal to (>=) 1 and Less Than (<) 1
Description: Percentage of participants with Th1 (IFN-g OR IL2 NOT TH2) /Th2 (IL4 OR IL5 OR IL13 AND CD40L) ratio >=1 and <1 was reported.
Time Frame: Days 15, 29, 57, 71, 85, 239 and 422
Population: as for outcome 55
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo
Number analyzed (Participants) | 27 | 29 | 30 | 28 | 6
Percentage of participants
  Day 15: Th1/Th2 >=1: number analyzed (Participants) | 27 | 29 | 29 | 28 | 3
  Day 15: Th1/Th2 >=1 | 100 [87 to 100] | 100 [88 to 100] | 100 [88 to 100] | 100 [88 to 100] | 100 [29 to 100]
  Day 15: Th1/Th2 <1: number analyzed (Participants) | 27 | 29 | 30 | 28 | 3
  Day 15: Th1/Th2 <1 | 0 [0 to 13] | 0 [0 to 12] | 0 [0 to 12] | 0 [0 to 12] | 0 [0 to 71]
  Day 29: Th1/Th2 >=1: number analyzed (Participants) | 27 | 25 | 28 | 23 | 6
  Day 29: Th1/Th2 >=1 | 100 [87 to 100] | 100 [86 to 100] | 100 [88 to 100] | 100 [85 to 100] | 100 [54 to 100]
  Day 29: Th1/Th2 <1: number analyzed (Participants) | 27 | 25 | 28 | 23 | 6
  Day 29: Th1/Th2 <1 | 0 [0 to 13] | 0 [0 to 14] | 0 [0 to 12] | 0 [0 to 15] | 0 [0 to 46]
  Day 57: Th1/Th2 >=1: number analyzed (Participants) | 27 | 19 | 27 | 19 | 4
  Day 57: Th1/Th2 >=1 | 100 [87 to 100] | 100 [82 to 100] | 100 [87 to 100] | 100 [82 to 100] | 100 [40 to 100]
  Day 57: Th1/Th2 <1: number analyzed (Participants) | 27 | 19 | 27 | 19 | 4
  Day 57: Th1/Th2 <1 | 0 [0 to 13] | 0 [0 to 18] | 0 [0 to 13] | 0 [0 to 18] | 0 [0 to 60]
  Day 71: Th1/Th2 >=1: number analyzed (Participants) | 22 | 17 | 30 | 17 | 4
  Day 71: Th1/Th2 >=1 | 100 [85 to 100] | 100 [80 to 100] | 100 [88 to 100] | 100 [80 to 100] | 100 [40 to 100]
  Day 71: Th1/Th2 <1: number analyzed (Participants) | 22 | 17 | 30 | 17 | 4
  Day 71: Th1/Th2 <1 | 0 [0 to 15] | 0 [0 to 20] | 0 [0 to 12] | 0 [0 to 20] | 0 [0 to 60]
  Day 85: Th1/Th2 >=1: number analyzed (Participants) | 25 | 15 | 28 | 16 | 4
  Day 85: Th1/Th2 >=1 | 100 [86 to 100] | 100 [78 to 100] | 100 [88 to 100] | 100 [79 to 100] | 100 [40 to 100]
  Day 85: Th1/Th2 <1: number analyzed (Participants) | 25 | 15 | 28 | 16 | 4
  Day 85: Th1/Th2 <1 | 0 [0 to 14] | 0 [0 to 22] | 0 [0 to 12] | 0 [0 to 21] | 0 [0 to 60]
  Day 239: Th1/Th2 >=1: number analyzed (Participants) | 15 | 16 | 9 | 4 | 0
  Day 239: Th1/Th2 >=1 | 100 [78 to 100] | 100 [79 to 100] | 100 [66 to 100] | 100 [40 to 100] |
  Day 239: Th1/Th2 <1: number analyzed (Participants) | 15 | 16 | 9 | 4 | 0
  Day 239: Th1/Th2 <1 | 0 [0 to 22] | 0 [0 to 21] | 0 [0 to 34] | 0 [0 to 60] |
  Day 422: Th1/Th2 >=1: number analyzed (Participants) | 6 | 10 | 7 | 4 | 0
  Day 422: Th1/Th2 >=1 | 86 [42 to 100] | 100 [69 to 100] | 100 [59 to 100] | 100 [40 to 100] |
  Day 422: Th1/Th2 <1: number analyzed (Participants) | 6 | 10 | 7 | 4 | 0
  Day 422: Th1/Th2 <1 | 14 [0 to 58] | 0 [0 to 31] | 0 [0 to 41] | 0 [0 to 60] |

68. Secondary Outcome: Cohort 2a: Percentage of Participants With T Helper Cell 1/T Helper Cell 2 Ratio (Th1/Th2) Greater Than or Equal to (>=) 1 and Less Than (<) 1
Description: as for outcome 67
Time Frame: Days 29 and 366
Population: PPI population was analyzed. Here, 'N' (Overall number of participants analyzed) =participants who were evaluable for this outcome measure and "n" (number analyzed) =participants who were evaluable for specified time points. Due to change in planned analysis, data was not collected and analyzed for "COHORT 2A: Placebo, B: PL" arm in this outcome measure. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: PL
Number analyzed (Participants) | 11 | 5 | 5 | 0
Percentage of participants
  Day 29: Th1/Th2 >=1: number analyzed (Participants) | 9 | 4 | 4 | 0
  Day 29: Th1/Th2 >=1 | 100 [66 to 100] | 100 [40 to 100] | 100 [40 to 100] |
  Day 29: Th1/Th2 <1: number analyzed (Participants) | 9 | 4 | 4 | 0
  Day 29: Th1/Th2 <1 | 0 [0 to 34] | 0 [0 to 60] | 0 [0 to 60] |
  Day 366: Th1/Th2 >=1: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 366: Th1/Th2 >=1 | 100 [3 to 100] | 100 [3 to 100] |  |
  Day 366: Th1/Th2 <1: number analyzed (Participants) | 1 | 1 | 0 | 0
  Day 366: Th1/Th2 <1 | 0 [0 to 98] | 0 [0 to 98] |  |

69. Secondary Outcome: Cohort 2b: Percentage of Participants With T Helper Cell 1/T Helper Cell 2 Ratio (Th1/Th2) Greater Than or Equal to (>=) 1 and Less Than (<) 1
Description: as for outcome 67
Time Frame: Days 29, 57, 85 and 422
Population: PPI population was analyzed. Here, 'N' (Overall number of participants analyzed) =participants who were evaluable for this outcome measure and "n" (number analyzed) =participants who were evaluable for specified time points. Due to change in planned analysis, data was not collected and analyzed for "COHORT 2B: Placebo, B: PL" arm in this outcome measure. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL
Number analyzed (Participants) | 12 | 5 | 6 | 0
Percentage of participants
  Day 29: Th1/Th2 >=1: number analyzed (Participants) | 9 | 2 | 3 | 0
  Day 29: Th1/Th2 >=1 | 100 [66 to 100] | 100 [16 to 100] | 100 [29 to 100] |
  Day 29: Th1/Th2 <1: number analyzed (Participants) | 9 | 2 | 3 | 0
  Day 29: Th1/Th2 <1 | 0 [0 to 34] | 0 [0 to 84] | 0 [0 to 71] |
  Day 57: Th1/Th2 >=1: number analyzed (Participants) | 9 | 4 | 1 | 0
  Day 57: Th1/Th2 >=1 | 100 [66 to 100] | 100 [40 to 100] | 100 [3 to 100] |
  Day 57: Th1/Th2 <1: number analyzed (Participants) | 9 | 4 | 1 | 0
  Day 57: Th1/Th2 <1 | 0 [0 to 34] | 0 [0 to 60] | 0 [0 to 98] |
  Day 85: Th1/Th2 >=1: number analyzed (Participants) | 6 | 4 | 3 | 0
  Day 85: Th1/Th2 >=1 | 100 [54 to 100] | 100 [40 to 100] | 100 [29 to 100] |
  Day 85: Th1/Th2 <1: number analyzed (Participants) | 6 | 4 | 3 | 0
  Day 85: Th1/Th2 <1 | 0 [0 to 46] | 0 [0 to 60] | 0 [0 to 71] |
  Day 422: Th1/Th2 >=1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 422: Th1/Th2 >=1 |  |  | 100 [3 to 100] |
  Day 422: Th1/Th2 <1: number analyzed (Participants) | 0 | 0 | 1 | 0
  Day 422: Th1/Th2 <1 |  |  | 0 [0 to 98] |

70. Secondary Outcome: Cohort 3: Percentage of Participants With T Helper Cell 1/T Helper Cell 2 Ratio (Th1/Th2) Greater Than or Equal to (>=) 1 and Less Than (<) 1
Description: Percentage of participant with Th1 (IFN-g OR IL2 NOT TH2) /Th2 (IL4 OR IL5 OR IL13 AND CD40L) ratio >=1 and <1 was reported.
Time Frame: Days 15, 29, 87, 100, 114 and 268
Population: FAS included all participant with at least one vaccine administration documented. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and "n" (number analyzed) signifies those participants who were evaluable for specified time points. "0" in the number analyzed field signifies that no participant was available for the analysis at the specified timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
Number analyzed (Participants) | 25 | 25 | 23 | 30 | 5
Percentage of participants
  Day 15: Th1/Th2 ratio >=1: number analyzed (Participants) | 23 | 22 | 22 | 24 | 2
  Day 15: Th1/Th2 ratio >=1 | 100 [85 to 100] | 100 [85 to 100] | 100 [85 to 100] | 100 [86 to 100] | 100 [16 to 100]
  Day 15: Th1/Th2 ratio <1: number analyzed (Participants) | 23 | 22 | 22 | 24 | 2
  Day 15: Th1/Th2 ratio <1 | 0 [0 to 15] | 0 [0 to 15] | 0 [0 to 15] | 0 [0 to 14] | 0 [0 to 84]
  Day 29: Th1/Th2 ratio >=1: number analyzed (Participants) | 25 | 25 | 23 | 30 | 4
  Day 29: Th1/Th2 ratio >=1 | 100 [86 to 100] | 100 [86 to 100] | 100 [85 to 100] | 100 [88 to 100] | 100 [40 to 100]
  Day 29: Th1/Th2 ratio <1: number analyzed (Participants) | 25 | 25 | 23 | 30 | 4
  Day 29: Th1/Th2 ratio <1 | 0 [0 to 14] | 0 [0 to 14] | 0 [0 to 15] | 0 [0 to 12] | 0 [0 to 60]
  Day 87: Th1/Th2 ratio >=1: number analyzed (Participants) | 13 | 12 | 9 | 17 | 1
  Day 87: Th1/Th2 ratio >=1 | 100 [75 to 100] | 100 [74 to 100] | 100 [66 to 100] | 100 [80 to 100] | 100 [3 to 100]
  Day 87: Th1/Th2 ratio <1: number analyzed (Participants) | 13 | 12 | 9 | 17 | 1
  Day 87: Th1/Th2 ratio <1 | 0 [0 to 25] | 0 [0 to 26] | 0 [0 to 34] | 0 [0 to 20] | 0 [0 to 98]
  Day 100: Th1/Th2 ratio >=1: number analyzed (Participants) | 20 | 19 | 21 | 21 | 1
  Day 100: Th1/Th2 ratio >=1 | 100 [83 to 100] | 100 [82 to 100] | 100 [84 to 100] | 100 [84 to 100] | 100 [3 to 100]
  Day 100: Th1/Th2 ratio <1: number analyzed (Participants) | 20 | 19 | 21 | 21 | 1
  Day 100: Th1/Th2 ratio <1 | 0 [0 to 17] | 0 [0 to 18] | 0 [0 to 16] | 0 [0 to 16] | 0 [0 to 98]
  Day 114: Th1/Th2 ratio >=1: number analyzed (Participants) | 24 | 20 | 20 | 16 | 5
  Day 114: Th1/Th2 ratio >=1 | 100 [86 to 100] | 100 [83 to 100] | 100 [83 to 100] | 100 [79 to 100] | 100 [48 to 100]
  Day 114: Th1/Th2 ratio <1: number analyzed (Participants) | 24 | 20 | 20 | 16 | 5
  Day 114: Th1/Th2 ratio <1 | 0 [0 to 14] | 0 [0 to 17] | 0 [0 to 17] | 0 [0 to 21] | 0 [0 to 52]
  Day 268: Th1/Th2 ratio >=1: number analyzed (Participants) | 16 | 17 | 4 | 8 | 0
  Day 268: Th1/Th2 ratio >=1 | 100 [79 to 100] | 94 [73 to 100] | 80 [28 to 99] | 89 [52 to 100] |
  Day 268: Th1/Th2 ratio <1: number analyzed (Participants) | 16 | 17 | 4 | 8 | 0
  Day 268: Th1/Th2 ratio <1 | 0 [0 to 21] | 6 [0 to 27] | 20 [1 to 72] | 11 [0 to 48] |

ADVERSE EVENTS:
Time Frame: Cohorts 1, 2a and 3: From Day 1 up to 808 days; Cohort 2b: Day 1 up to 752 days
Description: FAS included all subjects with at least one vaccine administration documented.
Groups:
- COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10): Healthy adult participants aged >=18 to <=55 received a single IM injection of Ad26.COV2.S 1*10^11 vp on Day 1 (Vaccination 1) and Day 57 (Vaccination 2). As per protocol amendment 15, all eligible participants who had previously received 1 or more doses of any COVID-19 vaccine were offered a single ad AHBV of Ad26.COV2.S at the dose of 5*10^10 vp Ad26.COV2.S. >=6 months after Vaccination 2.
- COHORT 2A: Placebo, B: Placebo: Group 5 subjects received a single IM injection of placebo matching to Ad26.COV2.S vaccine on Day 1 (Vaccination 1), 6 months (Booster 1) and 12 months (Booster 2). Subjects who had previously received 1 or more doses of any COVID-19 vaccine received a single ad hoc booster dose of 5*10^10 vp Ad26.COV2.S. 6 months after Booster 2 Vaccination.
Arm/Group | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1A: Placebo, Placebo | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 1B: Placebo, Placebo | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2A: Placebo, B: Placebo | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 | COHORT 2B: Placebo, B: PL | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) | COHORT 3: Placebo, Placebo
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/75 | 0/75 | 0/73 | 0/77 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/58 | 0/29 | 1/32 | 0/17 | 1/62 | 0/30 | 0/28 | 0/15 | 0/81 | 2/80 | 0/82 | 1/79 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/77 | 1/75 | 1/75 | 1/73 | 2/77 | 1/5 | 0/5 | 0/5 | 0/5 | 0/5 | 1/58 | 0/29 | 1/32 | 0/17 | 1/62 | 1/30 | 0/28 | 0/15 | 3/81 | 2/80 | 2/82 | 1/79 | 2/81
Other Adverse Events (participants affected / at risk) | 68/77 | 64/75 | 69/75 | 66/73 | 29/77 | 5/5 | 5/5 | 5/5 | 5/5 | 5/5 | 53/58 | 27/29 | 27/32 | 10/17 | 59/62 | 28/30 | 23/28 | 9/15 | 63/81 | 55/80 | 69/82 | 61/79 | 42/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) (N=77) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) (N=75) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) (N=75) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) (N=73) | COHORT 1A: Placebo, Placebo (N=77) | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Placebo, Placebo (N=5) | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) (N=58) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL (N=29) | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 (N=32) | COHORT 2A: Placebo, B: Placebo (N=17) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) (N=62) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL (N=30) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 (N=28) | COHORT 2B: Placebo, B: PL (N=15) | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) (N=81) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) (N=80) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) (N=82) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) (N=79) | COHORT 3: Placebo, Placebo (N=81)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aural Polyp (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hanging (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Legionella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple Sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1A: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) (N=77) | COHORT 1A: Ad26 5e10, PL(AHBV: Ad26 5e10) (N=75) | COHORT 1A: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) (N=75) | COHORT 1A: Ad26 1e11, PL(AHBV: Ad26 5e10) (N=73) | COHORT 1A: Placebo, Placebo (N=77) | COHORT 1B: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Ad26 5e10, PL(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Ad26 1e11, PL(AHBV: Ad26 5e10) (N=5) | COHORT 1B: Placebo, Placebo (N=5) | COHORT 2A: Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) (N=58) | COHORT 2A: Ad26 5e10, B: Ad26 5e10, PL (N=29) | COHORT 2A: Ad26 5e10, B: PL, Ad26 5e10 (N=32) | COHORT 2A: Placebo, B: Placebo (N=17) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL(PL/AHBV: Ad26 5e10) (N=62) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: Ad26 5e10, PL (N=30) | COHORT 2B: Ad26 5e10, Ad26 5e10, B: PL, Ad26 5e10 (N=28) | COHORT 2B: Placebo, B: PL (N=15) | COHORT 3: Ad26 5e10, Ad26 5e10(AHBV: Ad26 5e10) (N=81) | COHORT 3: Ad26 5e10, PL(AHBV: Ad26 5e10) (N=80) | COHORT 3: Ad26 1e11, Ad26 1e11(AHBV: Ad26 5e10) (N=82) | COHORT 3: Ad26 1e11, PL(AHBV: Ad26 5e10) (N=79) | COHORT 3: Placebo, Placebo (N=81)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea(Solicited) (Gastrointestinal disorders) | 19 (22) | 22 (27) | 25 (29) | 27 (31) | 5 (5) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 19 (19) | 8 (8) | 4 (4) | 2 (2) | 22 (27) | 8 (10) | 9 (10) | 2 (3) | 5 (5) | 7 (7) | 11 (11) | 9 (12) | 11 (11)
Chills (General disorders) | 3 (3) | 3 (3) | 6 (6) | 11 (11) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 6 (6) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (4) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Fatigue(Solicited) (General disorders) | 50 (72) | 41 (52) | 58 (89) | 53 (63) | 17 (21) | 4 (5) | 3 (4) | 5 (8) | 5 (6) | 4 (6) | 37 (37) | 17 (17) | 15 (15) | 7 (7) | 43 (67) | 15 (26) | 19 (30) | 4 (5) | 38 (49) | 32 (40) | 42 (59) | 39 (48) | 22 (29)
Injection Site Haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia(Solicited) (General disorders) | 13 (14) | 14 (14) | 33 (43) | 28 (29) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 15 (15) | 3 (3) | 4 (4) | 0 (0) | 17 (19) | 3 (4) | 6 (8) | 0 (0) | 5 (5) | 3 (3) | 7 (8) | 7 (7) | 1 (1)
Vaccination Site Erythema(Solicited) (General disorders) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Vaccination Site Pain(Solicited) (General disorders) | 58 (99) | 51 (55) | 64 (112) | 60 (66) | 9 (10) | 5 (8) | 3 (3) | 5 (10) | 4 (5) | 0 (0) | 48 (48) | 23 (23) | 19 (19) | 4 (4) | 53 (93) | 26 (44) | 20 (36) | 3 (3) | 50 (79) | 32 (34) | 55 (83) | 37 (45) | 14 (17)
Vaccination Site Swelling(Solicited) (General disorders) | 3 (4) | 0 (0) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Asymptomatic Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Lobe Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 31 (48) | 34 (37) | 52 (77) | 48 (51) | 4 (4) | 2 (3) | 3 (3) | 5 (7) | 5 (5) | 1 (1) | 34 (34) | 17 (17) | 13 (13) | 4 (4) | 32 (51) | 20 (27) | 16 (25) | 2 (2) | 26 (34) | 18 (23) | 35 (39) | 27 (31) | 12 (13)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 1 (1)
Headache(Solicited) (Nervous system disorders) | 41 (59) | 36 (48) | 52 (79) | 54 (64) | 14 (19) | 2 (3) | 3 (5) | 5 (9) | 5 (5) | 3 (3) | 35 (35) | 16 (16) | 11 (11) | 4 (4) | 43 (69) | 23 (30) | 18 (29) | 7 (8) | 32 (43) | 27 (32) | 39 (58) | 28 (41) | 21 (27)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine Spasm (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (3):
  • Study Protocol (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT04436276/Prot_001.pdf
  • Statistical Analysis Plan (2022-09-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT04436276/SAP_002.pdf
  • Informed Consent Form (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT04436276/ICF_003.pdf